CLINICAL TRIAL: NCT05934851
Title: A Prospective, Randomized, Single-blinded Study Evaluating the Effect of Frozen-Section Directed Excision on Positive Surgical Margins in High-grade Vulvar Dysplasia
Brief Title: A Study Evaluating the Effect of Frozen-Section Directed Excision Surgery on Vulvar Dysplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00094930; LCI-GYN-VUL-FSDE-001 (Other: Atrium Health); NCI-2024-03779 (Other: National Cancer Institute)
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Vulvar Neoplasm; Dysplasia Vulvar
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: After randomization, the surgical assignment will be revealed to the attending surgeon. Subjects will remain blinded until the six-month post-operative study visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frozen-Section Directed Excision Vulvectomy (Experimental): The surgeon(s) will identify the lesion and make a 1 mm excision around the lesion site.
  Interventions: Procedure: Frozen-Section Directed Excision
- Wide Local Excision Vulvectomy (Active Comparator): The surgeon(s) will visually identify the abnormal lesion. A Wide Local Excision with 5 mm margins will be made through the dermis per standard of care.
  Interventions: Procedure: Wide Local Excision

INTERVENTIONS:
Procedure: Frozen-Section Directed Excision — Frozen-Section Directed Excision (FSDE) is a surgical technique with evaluation of margin status during the surgical procedure, similar to the established Mohs Surgical Technique. The use of FSDE may ensure negative margins, decrease unnecessary excision of healthy tissue and has the potential to greatly reduce positive margins.
  Other Names: FSDE
  Arms: Frozen-Section Directed Excision Vulvectomy
Procedure: Wide Local Excision — Standard of care surgical technique utilized for VIN 2, VIN3, VIN 2/3 or High-grade Dysplasia NOS
  Arms: Wide Local Excision Vulvectomy

SUMMARY:
The purpose of this study is to compare "Frozen-Section Directed Excision", which has been a proven method of surgery used in dermatology, versus the current, standard method called "Wide Local Excision" to treat high-grade vulvar dysplasia.

DETAILED DESCRIPTION:
This is a randomized, single-blinded study. The target population is adults ≥ 18 years of age with histological or cytological confirmation of VIN 2, VIN 3, VIN 2/3 or High-grade Dysplasia NOS with a planned excisional procedure, with high suspicion by the enrolling investigator that gross surgical margins of ≥ 3 mm can be achieved without laser or other destructive procedures. One group of subjects will be assigned to the Frozen-Section Directed Excision surgery arm and will undergo this procedure. The other group of subjects will be assigned to the Wide Local Excision (standard of care) arm and will undergo this procedure. The randomization will be 1:1, meaning for every subject who gets assigned to the Frozen-Section Directed Excision surgery arm, one will also be assigned to the Wide Local Excision arm. There is a 50% chance of getting randomized to either the Frozen-Section Directed Excision procedure or Wide Local Excision. Information regarding the surgery procedure, the amount of time the surgery procedure takes, and total amount of pain medication required during surgery and while in the surgery recovery area will be collected. The study team will also look at recurrence rates (return of the cancer) in six months, if any other therapies are required, and subject satisfaction related to the surgery, recovery, and sexual function by using questionnaires before and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information.
2. Age ≥ 18 years at the time of consent
3. Histological or cytological confirmation of VIN 2, VIN 3, VIN 2/3 or High-grade Dysplasia NOS with a planned excisional procedure, with high suspicion by the enrolling investigator that gross surgical margins of ≥ 3 mm can be achieved without laser or other destructive procedures
4. Surgery is expected to occur within 90 days from randomization
5. Ability to read and understand the English and/or Spanish language
6. As determined by the enrolling physician, ability and willingness of the subject to comply with study procedures for the entire length of the study
7. No known pregnancy

Exclusion Criteria:

1. Excision is not possible due to anatomy (proximity to urethra/clitoris)
2. Known immunodeficiency syndrome
3. Immunosuppressant medications taken within the last 30 days (HIV, organ transplant recipient, chronic steroid use/immunosuppressant)
4. History of pelvic region radiation therapy
5. Active anticancer treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Rates of positive margins for VIN 2, VIN 3, VIN 2/3 or High-grade Dysplasia NOS | At the time of the resection
  Comparison of rates of positive margins for VIN 2, VIN 3, VIN 2/3 or High-grade Dysplasia NOS in subjects who undergo standard of care Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision

SECONDARY OUTCOMES:
Recurrence rates at 6 months | 6 months post resection surgery
  Comparison of recurrence rates in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision
Surgical time | At the time of the resection
  Comparison of surgical time in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision
Recovery room time | At the time of the resection and recovery
  Comparison of recovery room time in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision
Narcotic dose required (total during surgery and in recovery) | At the time of the resection and recovery
  Comparison of narcotic dose required in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision
Blood loss | At the time of the resection
  Comparison of blood loss in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision
Primary wound closure rates | 2-week post resection surgery
  Comparison of primary wound closure rates in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision
Post-operative quality of life as determined by the SSQ-8 | 2-weeks and 6 months after resection surgery
  Comparison of post-operative quality of life as determined by the SSQ-8 in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision
Sexual function as determined by the FSFI | Screening and 6 months after resection surgery
  Comparison of sexual function as determined by the FSFI in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision
Wound bed size after surgery | End of resection surgery
  Comparison of wound bed size after surgery in subjects who undergo standard Wide Local Excision versus subjects who undergo Frozen-Section Directed Excision

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Naumann, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No